CLINICAL TRIAL: NCT03663621
Title: How to Reach Women of Reproductive Age With Obesity to Support Weight Loss Before Pregnancy?
Brief Title: Prepare - How to Reach Women of Reproductive Age With Obesity to Support Weight Loss Before Pregnancy?
Status: Completed | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1105007
Record Dates: First submitted 2018-03-01; First posted 2018-09-10 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Pregnancy Complications
MeSH Terms: conditions — Obesity; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initial survey and interview (Aim 2): Participants in Aim 2 will be asked to complete an initial 15-minute survey and 20-30 minute semi-structured interview. The purpose of this study is to learn the best ways to support healthful behaviors and weight loss prior to pregnancy. Researchers are also interested in what motivates or prevents women of reproductive age from engaging in a structured weight loss program.
- Formal weight loss program (Aim 3): Participants in Aim 3 have expressed interest in referral to the Mass General Weight Center. The purpose of this study is to learn what motivates or prevents women of reproductive age from engaging in a structured weight loss program. Researchers will ask for no more than a half hour of participant's time to complete a 5- minute interview following Orientation at the Weight Center and another 10-minute interview after a participant has participated in a program offered at the Weight Center.

SUMMARY:
Researchers at Harvard Pilgrim Health Care Institute and Massachusetts General Hospital are conducting a study to learn more about how best to reach out to women (age 18-45) who are thinking about a pregnancy in the next couple of years and currently have a BMI greater than 30 kg/m2.

Interested participants will be asked to complete a 15-minute survey. The survey will ask some more questions about their prior reproductive health history, opinions and experiences regarding lifestyle, weight and health. After completing the survey, researchers would like to arrange a time to complete a 20- to 30-minute semi-structured interview about their perceived health in the process of planning pregnancy.

DETAILED DESCRIPTION:
The purpose of this study is to learn the best ways to support healthful behaviors and weight loss prior to pregnancy. Researchers are also interested in what motivates or prevents women of reproductive age from engaging in a structured weight loss program. Participants will be asked for no more than an hour of their time to complete a brief survey and participate in an interview. This study is being conducted by Harvard Pilgrim Health Care Institute. This study is being paid for by the Nutrition Obesity Research Center at Harvard (NORCH).

At the end of the interview, study staff will also talk to participants about the opportunity to be referred to the Mass General Weight Center if they are interested in participating in a program now being offered there.

If participants elect to participate in a program at the weight center, researchers would then like to complete 2 more short interviews with these participants about that process. The first will be about 5 minutes and will take place just after the initial Weight Center Orientation, and the last will be about 10 minutes and take place after 3 months of participation. During this final interview, researchers will ask for participant opinions about the program that they have just participated in.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years old,
* BMI>30 mg/m2,
* thinking about planning a pregnancy in the next 2 years

Exclusion Criteria:

* Previous bariatric surgery,
* currently pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will include patients in Massachusetts General Hospital clinical settings, users of the Ovia fertility app as well as members of the community who may see ads posted in local newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Participant recruitment feasibility | 1 year
  Feasibility determined by compiling the actual number of participants recruited divided by the time and resources necessary to achieve that number participants for each recruitment strategy.

SECONDARY OUTCOMES:
Participants' attitudes and perceptions of their own health risks with regard to weight-related complications | 1 year
  Participants are asked to measure levels of agreement/disagreement with their perceived health risk for ten weight related complications as follows: developing developing diabetes, developing cancer, developing heart disease, developing high blood pressure, developing high cholesterol, being able to get pregnant, having diabetes during pregnancy, having high blood pressure during pregnancy, having a large baby, and having to undergo a c-section
Participant adherence during a structured weight loss program. | 1 year
  Participants' attendance is recorded throughout the duration of a 12-week weight loss program. Successful adherents will have attended >70% of meetings.
Participants' estimated time frame before trying to get pregnant and willingness to delay their pregnancy attempt in order to complete a structured weight loss program. | 1 year
  Participants are interviewed to assess their current time frame before actively trying to get pregnant. Participants are also asked if they are willing to delay a pregnancy attempt and if so, for how long.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Hivert, MD, MMSc, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Harvard Pilgrim Health Care Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No